CLINICAL TRIAL: NCT06624800
Title: The Efficacy and Safety of Shoulder Chuna on in Patients with Shoulder Pain Caused by Traffic Accidents: a Pragmatic Randomized Controlled Trial
Brief Title: The Efficacy and Safety of Shoulder Chuna on in Patients with Shoulder Pain Caused by Traffic Accidents
Acronym: Shoulder chuna
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JS-CT-2024-08; Jaseng Medical Foundation (Other: Jaseng Medical Foundation)
Record Dates: First submitted 2024-09-26; First posted 2024-10-03 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Acute Shoulder Pain
Keywords: shoulder chuna therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Shoulder chuna treatment (Experimental): During the hospitalization period, Chuna therapy for the shoulder joint will be performed once a day for a total of 10 to 15 minutes, including before, during, and after the treatment. The practitioner will assess the condition and select one of three techniques-posterior displacement, anterior displacement, or lateral displacement-to apply Chuna therapy
  Interventions: Procedure: Korean medical treatment
- Korean medical treatment (Active Comparator): The control group were received Korean medical treatment everyday after hospitalization: acupuncture, chuna, pharmacoacupuncture and Korean herbal medicine.
  Interventions: Procedure: Shoulder chuna treatment(posterior displacement, anterior displacement, or lateral displacement); Procedure: Korean medical treatment

INTERVENTIONS:
Procedure: Shoulder chuna treatment(posterior displacement, anterior displacement, or lateral displacement) — The Shoulder Chuna therapy for the shoulder joint will be performed on the affected shoulder from the second day of hospitalization until the day before discharge.
  Arms: Korean medical treatment
Procedure: Korean medical treatment — acupuncture treatment, chuna, pharmacoacupuncture, Korean herbal medicine

SUMMARY:
This study is a double blind, randomized controlled trail. condition/disease: Patient with acute shoulder pain and restricted movement due to a traffic accident. treatment/intervention: Chuna therapy for the shoulder, including integrated Korean medicine treatment

DETAILED DESCRIPTION:
The investigators intend to conduct a randomized controlled trial to evaluate the effectiveness of Chuna therapy for shoulder pain and restricted movement caused by a traffic accident. The study will involve administering shoulder Chuna therapy from the second day of hospitalization until discharge, with the aim of assessing its effects on shoulder pain relief and recovery of range of motion. Although the effectiveness of Korean medicine for treating trauma from traffic accidents has been well studied, the research has largely focused on spinal conditions, such as those affecting the cervical and lumbar spine. Likewise, most studies on Chuna therapy have centered around spinal disorders. Through this study, the investigators aim to explore the therapeutic effects of shoulder Chuna therapy, an area that has not been extensively researched.

1. The effectiveness of shoulder Chuna therapy will be evaluated by observing and comparing changes in pain, range of motion limitation, functional disability, quality of life, and patient satisfaction between the shoulder Chuna group (treatment group) and the Korean integrative medicine group (control group).
2. Investigators will assess the treatment effects of shoulder Chuna therapy on shoulder pain and restricted movement by observing improvements in initial NRS, VAS scores, SPADI, and ROM in the shoulder Chuna group (treatment group) compared to the Korean integrative medicine group (control group).
3. The total number of treatment sessions and the degree of improvement will be observed and compared between the shoulder Chuna group (treatment group) and the Korean integrative medicine group (control group) to evaluate the effectiveness of the treatment frequency.
4. The safety of the therapy will be assessed by investigating adverse reactions in both the shoulder Chuna group (treatment group) and the Korean integrative medicine group (control group).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 19-69 years on the date they sign the consent form.
* Patients with shoulder pain and restricted movement occurring within 5 days after a traffic accident.
* Patients who are hospitalized due to traffic accident.
* Patients with NRS of shoulder pain ≥ 5 with restricted movement due to a traffic accident.
* Patients who provide consent to participate in the trial and return the informed consent form.

Exclusion Criteria:

* Patients with a specific serious disease that may cause shoulder pain: malignancy, spondylitis, inflammatory spondylitis, etc.
* Patients with progressive neurological deficits or with severe neurological symptoms.
* Patients with medical history of cervical surgery or shoulder surgery within the last three weeks.
* Patients with a specific serious disease that may interfere with the interpretation of the therapeutic effects or results: malignancy, spondylitis, inflammatory spondylitis, etc.
* Chuna therapy is deemed inappropriate or unsafe due to conditions like fractures, dislocations, ligament tears, or unstable healing fractures; skeletal demineralization and ligament laxity with subluxation or dislocation; or inflammation
* Presence of other chronic diseases that could interfere with treatment outcomes or interpretation, such as cardiovascular disease, kidney disease, diabetic neuropathy, dementia, or epilepsy
* Currently taking steroids, immunosuppressants, psychiatric medications, or other drugs that may affect study results
* Acupuncture is deemed inappropriate or unsafe, such as in patients with bleeding disorders, those on anticoagulant therapy, those with severe diabetes prone to infection, or those with severe cardiovascular disease
* Patients who are pregnant or planning to become pregnant.
* Patients who are presence of severe mental illness
* Patients who are participated in clinical trials other than observational studies without therapeutic intervention.
* Patients who are difficult to complete the research participation agreement.
* Other patients whose participation in the trial is judged by a researcher to be problematic.

Ages: 19 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale(NRS) of Shoulder pain | Screening, From baseline(Day2) up to Discharge 1 day, 2week after enrollment, 1month after enrollment, 3month after enrollment
  NRS is a pain scale in which the patient indicates their subjective pain as a whole number from 0 to 10. The participant is asked to report their shoulder pain and discomfort using NRS, where 0 indicates 'no pain or discomfort' and 10 indicates 'the most severe pain and discomfort imaginable'.

SECONDARY OUTCOMES:
Location of shoulder joint displacement | Screening, From baseline(Day2) up to Discharge 1 day, 2week after enrollment, 1month after enrollment, 3month after enrollment
  The location of shoulder pain varies depending on the nerve. The assessor will ask patients where the pain occur.
Shoulder Pain intensity scale: Visual Analogue Scale (VAS) | From baseline(Day2) up to Discharge 1 day
  VAS is an assessment index in which the patient records their pain on a 100mm line from 'no pain' at one end, and 'the most severe pain imaginable' at the other end.
Physical examination (Shoulder active range of motion) | From baseline(Day2) up to Discharge 1 day
  The patient's maximum active and passive range of motion (ROM) of the shoulder, which they can move without pain, will be measured. The shoulder ROM will include six movements: flexion, extension, adduction, abduction, internal rotation, and external rotation. Measurements will be taken before and after treatment using a goniometer. If the patient refuses the measurement due to severe pain or other reasons, a value of 0 degrees will be recorded.
Shoulder Pain and Disability Index(SPADI) | From baseline(Day2) up to Discharge 1 day, 2week after enrollment, 1month after enrollment, 3month after enrollment
  The patient's functional status will be assessed using the SPADI questionnaire. The SPADI was developed to evaluate the degree of disability related to shoulder pain and consists of 13 items in total: 5 items on the severity of pain and 8 items on the degree of discomfort. Each item is rated on a 10-point scale, with scores ranging from 0 to 10. Higher scores indicate greater disability. A validated Korean version of the SPADI questionnaire will be used.
EuroQol 5-Dimension (EQ-5D) | From baseline(Day2) up to Discharge 1 day, 2week after enrollment, 1month after enrollment, 3month after enrollment
  The EQ-5D is a method of indirectly calculating the weights of certain health states for quality of life after a multidimensional investigation of health states, and is the most widely used instrument for this purpose. The EQ-5D consists of 5 questions about current health state (mobility, self-care, usual activities, pain, anxiety/depression), and each question is scored on a 5-point Likert scale (1=no problems, 3=moderate problems, 5=severe problems). In this study, the investigators will use the Korean version of the EQ-5D, which has been demonstrated to be valid.
Patient Global Impression of Change (PGIC) | Discharge 1 day, 2week after enrollment, 1month after enrollment, 3month after enrollment
  The PGIC is an index that assesses improvements in functional limitation caused by whiplash injury. Participants rate the improvement in functional limitations after treatment on a 7-point Likert scale (1=Very much improved, 4=No change, 7=Very much worse). This index was originally developed for use in Psychology, but is currently used in various other medical fields to assess improvements in pain.

CONTACTS AND LOCATIONS:
Overall Officials: In-Hyuk Ha, phD, Study Director — Jaseng Medical Foundation
Locations (1):
- Jaseng Hospital of Korean Medicine, Seoul, Gangnam-Gu, South Korea

IPD SHARING:
Plan to Share IPD: No